CLINICAL TRIAL: NCT04652986
Title: Mid- and Long-term Surgical and Oncological Outcomes of Total Laparoscopic Gastrectomy for Gastric Cancer: A Prospective Study
Brief Title: Outcomes of Laparoscopic Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Juan Carlos Martín del Olmo (Other)
Responsible Party: Sponsor-Investigator, Juan Carlos Martín del Olmo, MD, PhD. Associate Professor Valladolid University., Hospital Medina del Campo
Organization: Hospital Medina del Campo (Other)
Other Study IDs: HMCampo
Record Dates: First submitted 2020-11-18; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Gastric Cancer; Laparoscopic Gastrectomy
Keywords: Gastric cancer; Laparoscopy; Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A prospective study of the results of laparoscopic approach of gastric carcinoma in western patients is designed. The working hypothesis proposes obtaining similar results to those obtained in the series reported by eastern hospitals (Japan and Korea) and, at least, equivalent to those recorded in conventional surgery.

DETAILED DESCRIPTION:
This is a single-center prospective study. All gastric adenocarcinoma patients operated on between January 2004 and December 2022 who underwent laparoscopic resection with D1-D2 lymphadenectomy were considered.

The exclusion criteria were patients who were lost to follow-up, were unfit for surgery, underwent palliative surgery or had T4b lesions or gastric neoplasms other than adenocarcinoma.

The preoperative evaluation included laboratory tests, upper digestive endoscopy with biopsy, computed tomography scans (chest, abdomen, and pelvis), and endoscopic ultrasound in selected cases.

The tumor node, metastasis (TNM) protocol of the College of American Pathologists was used for staging In the preoperative workup, the patients were classified according to the American Anesthesiology Association (ASA).

Perioperative and postoperative complications will be classified according to the Clavien-Dindo system.

Length of hospital stay, age, sex, comorbidities, extent of surgery, pTNM stage, and disease-free survival (DFS) will be analyzed.

The followed-up it is planned at one, three and six months after surgery and every 6 months later until the fifth year, then once a year.

Statistical analyses were performed using SPSS, ver. 25.0 (SPSS Inc., Chicago IL, USA). The demographics, perioperative data, operation details, length of hospital stay, morbidity, mortality and pathologic and oncological outcomes are expressed as numbers and percentages for qualitative variables and medians and interquartile ranges (IQRs) for quantitative variables.

Factors associated with recurrence risk at 12, 36 and 60 months will be evaluated using univariate and multivariate Cox regression analyses. Variables with P < 0.1 in the univariate analysis were further introduced into the multivariate analysis using the Wald selection method. TNM stage will be analyzed for its impact on DFS using the Kaplan-Meier method and the log-rank test at 12, 36 and 60 months.

To determine the risk factors for the development of serious morbidity (Clavien-Dindo ≥III), we first performed univariate and multivariate logistic regression analyses. Variables with P<0.1 in the univariate analysis will be further introduced into the multivariate analysis with the Wald selection method. P values < 0.05 were considered statistically significant.

This study involved the use of data from clinical records. To guarantee the proper handling of the information, the data were treated confidentially and anonymously according to the provisions of the Spanish Organic Law 15/1999, of 13 December 1999, on Personal Data Protection (LOPD). All methods were performed in accordance with the guidelines and regulations established by the Declaration of Helsinki (1964, revised in 1983) on biomedical research in humans, the Spanish Royal Decree 1090/2015, of December 4, which regulates clinical trials with drugs, the Research Ethics Committees with drugs and the Spanish Registry of Clinical Studies.

Ethical approval from the Clinical Trials and Ethics Committee of Valladolid University was granted.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of gastric adenocarcinoma fit for surgical treatment.

Exclusion Criteria:

* patients who were lost to follow-up
* patients unfit for surgery
* palliative surgery
* T4b lesions
* neoplasms other than adenocarcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed of gastric adenocarcinoma in the area care of Medina del Campo Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2004-01 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival at three years | Three years.
  Rate of patients who reach this condition
Disease-free survival at five years | Five years
  Rate of patients who reach this condition

SECONDARY OUTCOMES:
Three years overall survival | Three years.
  Rate of patients who reach this condition
Five years overall survival | Five years
  Rate of patients who reach this condition

OTHER OUTCOMES:
Operative mortality | One month
  Rate of patients died in the first thirty days
Operative morbidity | One month
  Rate of operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Martín del Olmo, MD,PhD, Study Director — Hospital de Medina del Campo
Locations (1):
- Juan Carlos Martín del Olmo, Medina del Campo, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suda K, Nakauchi M, Inaba K, Ishida Y, Uyama I. Minimally invasive surgery for upper gastrointestinal cancer: Our experience and review of the literature. World J Gastroenterol. 2016 May 21;22(19):4626-37. doi: 10.3748/wjg.v22.i19.4626. PMID 27217695
- [Background] Best LM, Mughal M, Gurusamy KS. Laparoscopic versus open gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2016 Mar 31;3(3):CD011389. doi: 10.1002/14651858.CD011389.pub2. PMID 27030300
- [Background] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- [Background] Li Z, Li B, Bai B, Yu P, Lian B, Zhao Q. Long-term outcomes of laparoscopic versus open D2 gastrectomy for advanced gastric cancer. Surg Oncol. 2018 Sep;27(3):441-448. doi: 10.1016/j.suronc.2018.05.022. Epub 2018 May 26. PMID 30217300
- [Background] Sano T, Sasako M, Yamamoto S, Nashimoto A, Kurita A, Hiratsuka M, Tsujinaka T, Kinoshita T, Arai K, Yamamura Y, Okajima K. Gastric cancer surgery: morbidity and mortality results from a prospective randomized controlled trial comparing D2 and extended para-aortic lymphadenectomy--Japan Clinical Oncology Group study 9501. J Clin Oncol. 2004 Jul 15;22(14):2767-73. doi: 10.1200/JCO.2004.10.184. Epub 2004 Jun 15. PMID 15199090
- [Background] Hendriksen BS, Brooks AJ, Hollenbeak CS, Taylor MD, Reed MF, Soybel DI. The Impact of Minimally Invasive Gastrectomy on Survival in the USA. J Gastrointest Surg. 2020 May;24(5):1000-1009. doi: 10.1007/s11605-019-04263-4. Epub 2019 May 31. PMID 31152343
- [Background] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Background] Lin JX, Lin JP, Desiderio J, Xie JW, Gemini A, Wang JB, Lu J, Chen QY, Cao LL, Lin M, Tu R, Zheng CH, Li P, Parisi A, Huang CM. Difference in the short-term outcomes of laparoscopic gastrectomy for gastric carcinoma between the east and west: a retrospective study from the IMIGASTRIC trial. J Cancer. 2019 Jul 10;10(17):4106-4113. doi: 10.7150/jca.31192. eCollection 2019. PMID 31417655
- [Background] Maida P, Marte G, Spedicato GA, Ferronetti A, Mauriello C, Canfora A, Ciorra G, Barra L, Di Maio V. Laparoscopic versus open gastrectomy with extended lymph node dissection for gastric carcinoma in a Western series: a Propensity Score Matching analysis. Minerva Chir. 2019 Feb;74(1):107-111. doi: 10.23736/S0026-4733.18.07562-4. No abstract available. PMID 30646677
- [Background] Treitl D, Hochwald SN, Bao PQ, Unger JM, Ben-David K. Laparoscopic Total Gastrectomy with D2 Lymphadenectomy and Side-to-Side Stapled Esophagojejunostomy. J Gastrointest Surg. 2016 Aug;20(8):1523-9. doi: 10.1007/s11605-016-3162-7. Epub 2016 May 16. PMID 27184675
- [Background] Guideline Committee of the Korean Gastric Cancer Association (KGCA), Development Working Group & Review Panel. Korean Practice Guideline for Gastric Cancer 2018: an Evidence-based, Multi-disciplinary Approach. J Gastric Cancer. 2019 Mar;19(1):1-48. doi: 10.5230/jgc.2019.19.e8. Epub 2019 Mar 19. No abstract available. PMID 30944757
- [Background] Yamamoto M, Shimokawa M, Kawano H, Ohta M, Yoshida D, Minami K, Ikebe M, Morita M, Toh Y. Benefits of laparoscopic surgery compared to open standard surgery for gastric carcinoma in elderly patients: propensity score-matching analysis. Surg Endosc. 2019 Feb;33(2):510-519. doi: 10.1007/s00464-018-6325-7. Epub 2018 Jul 20. PMID 30030615
- [Background] Kim W, Kim HH, Han SU, Kim MC, Hyung WJ, Ryu SW, Cho GS, Kim CY, Yang HK, Park DJ, Song KY, Lee SI, Ryu SY, Lee JH, Lee HJ; Korean Laparo-endoscopic Gastrointestinal Surgery Study (KLASS) Group. Decreased Morbidity of Laparoscopic Distal Gastrectomy Compared With Open Distal Gastrectomy for Stage I Gastric Cancer: Short-term Outcomes From a Multicenter Randomized Controlled Trial (KLASS-01). Ann Surg. 2016 Jan;263(1):28-35. doi: 10.1097/SLA.0000000000001346. PMID 26352529
- [Background] Shi Y, Xu X, Zhao Y, Qian F, Tang B, Hao Y, Luo H, Chen J, Yu P. Long-term oncologic outcomes of a randomized controlled trial comparing laparoscopic versus open gastrectomy with D2 lymph node dissection for advanced gastric cancer. Surgery. 2019 Jun;165(6):1211-1216. doi: 10.1016/j.surg.2019.01.003. Epub 2019 Feb 14. PMID 30772006
- [Background] Shimada S, Sawada N, Oae S, Seki J, Takano Y, Ishiyama Y, Nakahara K, Maeda C, Hidaka E, Ishida F, Kudo SE. Safety and curability of laparoscopic gastrectomy in elderly patients with gastric cancer. Surg Endosc. 2018 Oct;32(10):4277-4283. doi: 10.1007/s00464-018-6177-1. Epub 2018 Mar 30. PMID 29602987

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT04652986/Prot_SAP_000.pdf